CLINICAL TRIAL: NCT04613128
Title: A Prospective Study to Evaluate Biological and Clinical Effects of Significantly Corrected CFTR Function (the PROMISE Pediatric 6 to 11 Years Old Study)
Brief Title: The PROMISE Pediatric Study 6 to 11 Years Old
Status: Active, not recruiting | Type: Observational
Sponsor: Nicole Hamblett (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor-Investigator, Nicole Hamblett, Professor of Pediatrics, Division of Pulmonary and Sleep Medicine, University of Washington School of Medicine Adjunct Professor, Biostatistics, University of Washington School of Medicine Co-Executive Director, Cystic Fibrosis Therapeutics Development, Seattle Children's Hospital
Organization: Seattle Children's Hospital (Other)
Other Study IDs: PROMISE-OB-18 Pediatric Study
Record Dates: First submitted 2020-10-27; First posted 2020-11-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Cystic Fibrosis; Cystic Fibrosis in Children
Keywords: CF; Cystic Fibrosis; CFTR Modulator; Trikafta; Triple Combination Therapy; Pediatric; ETI; elexacaftor/texacaftor/ivacaftor
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, buffy coat, urine, sputum, oropharyngeal swab (throat swab), stool, sweat
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric: Cystic Fibrosis pediatric patients (6-11 years old) prescribed ETI CFTR modulator Therapy.

SUMMARY:
This is a prospective, multi-center observational study. The study is designed to measure the clinical effectiveness of elexacaftor, tezacaftor and ivacaftor (ETI) triple combination therapy in children (6-11 years of old) with one or more copies of the F508del mutation, study the effects of ETI across a number of CF disease manifestations, and collect specimens for future research. Subjects in the study will have one "before ETI" visit within 30 days before initiation of the therapy and five "after ETI" visits over a 24-month follow-up period. Participants who have participated in the original PROMISE Pediatric Sub-Study have the option of participating in a long-term extension with annual visits performed at the 36- and 48-month timepoints. The durability of the clinical and biological changes in the PROMISE Pediatric Sub-Study can be assessed with extended follow-up, which would enable the sub-studies to consider potential clinical consequences of the biological or physiological effects being studied. This work will help to inform long term prognosis and feasibility of certain clinical trials outcomes for interventional studies and may be useful when considering research priorities in drug development. The duration of participation for each subject is 24 months (with an additional 24 months if participants agree to the optional long-term extension). NOTE: FDA has granted approval for elexacaftor, tezacaftor and ivacaftor in the 6-11 age group.

DETAILED DESCRIPTION:
While nearly 2000 mutations have been described, the most common disease causing CFTR mutation is F508del, which is found in >85% of patients followed in the US CF Patient Registry. Two CFTR corrector drugs (elexacaftor and tezacaftor) plus the potentiator ivacaftor have been developed and approved as a triple combination therapy for CF patients (12 years old and above) with one or two copies of the F508del mutation. We predict that over 90% of pediatric CF patients (age 6-11 y/o) will be eligible for highly effective CFTR modulator therapy in the U.S.

The PROMISE Pediatric Study is designed to measure the direct and indirect CFTR dependent anion secretion by collecting and analyzing clinical research outcomes and biomarkers on pediatric patients both before and after they begin treatment with ETI. This study will investigate the impact of ETI across a wide range of CF disease manifestations and organ systems. While specific biomarkers of special interest have been selected for detailed analysis in this study, an additional important goal is to collect blood, urine, stool, and airway epithelial cell specimens for long-term storage in a biorepository to enable future research. These samples can be made available for research beyond the current scope of work. The PROMISE Pediatric Study will provide a coordinated collection of clinical research outcomes data that can be linked with these specimens.

ELIGIBILITY:
Inclusion Criteria:

1. Written parental informed consent and assent obtained from subject and the subject's legal guardian.
2. Be willing and able to adhere to the study visit schedule and other protocol requirements.
3. All genders 6-11 years old on Day 1.
4. Diagnosis of CF.
5. CFTR mutations consistent with the FDA labeled indication for the ETI.
6. Physician intent to prescribe the ETI.
7. Able to attempt the testing and procedures required for this study, as judged by the investigator.
8. Enrolled in the Cystic Fibrosis Foundation Patient Registry.
9. Clinically stable with no significant changes in health status within the 14 days prior to Visit 1 (and inclusive of Visit 1).

Exclusion Criteria:

1. Has any other condition that, in the opinion of the Site Investigator/designee, would preclude informed consent or assent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.
2. Use of any ETI within the 180 days prior to Visit 1.
3. Any acute use of antibiotics (oral, inhaled or IV) or acute use of systemic corticosteroids within the 14 days prior to Visit 1 (inclusive of Visit 1) for lower respiratory tract symptoms.
4. Initiation of any new chronic therapy (e.g., ibuprofen, Pulmozyme®, hypertonic saline, azithromycin, inhaled tobramycin, Cayston®, Kalydeco, Orkambi®, Symdeko®) within the 4 weeks prior to Visit 1 (inclusive of Visit 1).
5. Use of an investigational agent within the 28 days prior to Visit 1.
6. Use of chronic oral corticosteroids (equivalent to 10 mg. or more per day of prednisone) within the 28 days prior to Visit 1.
7. Treatment for nontuberculous mycobacterial (NTM) infection, consisting of ≥ two antibiotics (oral, IV, and/or inhaled) within the 28 days prior to Visit 1.
8. History of lung or liver transplantation,or listing for organ transplantation.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Cystic Fibrosis, 6-11 years old prescribed ETI.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2021-06-11 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Sweat Chloride at 6 months | 6 months
  Change in sweat chloride from Baseline to 6 months.
Sweat Chloride at 24 months | 24 months
  Change sweat chloride from Baseline to 24 months.
Forced expiratory volume at one second (FEV1) at 6 months | 6 months
  Change in FEV1 from Baseline to 6 months.
Forced expiratory volume at one second (FEV1) at 24 months | 24 months
  Change in FEV1 from Baseline to 24 months.
Lung Clearance Index (LCI) at 6 months | 6 months
  Change Lung Clearance Index (LCI) from baseline to 6 months.
Lung Clearance Index (LCI) at 24 months | 24 months
  Change Lung Clearance Index (LCI) from baseline to 24 months.

SECONDARY OUTCOMES:
Weight at 6 Months | 6 months
  Change in weight from Baseline to 6 months.
Weight at 24 Months | 24 months
  Change in weight from Baseline to 24 months.
BMI at 6 Months | 6 months
  Change in BMI from Baseline to 6 months.
BMI at 24 Months | 24 months
  Change in BMI from Baseline to 24 months.
Cystic Fibrosis Questionnaire Revised (CFQ-R) at 6 Months | 6 months
  Change in CFQ-R (respiratory domain) from Baseline to 6 months.
Cystic Fibrosis Questionnaire Revised (CFQ-R) at 24 Months | 24 months
  Change in CFQ-R (respiratory domain) from Baseline to 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Rowe, MD, Principal Investigator — University of Alabama at Birmingham; David Nichols, MD, Principal Investigator — University of Washington
Locations (20):
- United States (20):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University Medical Center, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - John Hopkins University, Baltimore, Maryland
  - Boston Children's Hospital, Brigham & Women's Hospital, Boston, Massachusetts
  - The Minnesota Cystic Fibrosis Center, Minneapolis, Minnesota
  - Children's Mercy Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital/University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Baylor College of Medicine, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No